CLINICAL TRIAL: NCT04198038
Title: A Pilot Study to Evaluate the Feasibility of Family-Centered Songwriting in Pediatric Palliative Care
Brief Title: Family-Centered Songwriting in Pediatric Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Terrah Akard, Associate Professor, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 191557
Record Dates: First submitted 2019-12-05; First posted 2019-12-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Cognitive Impairment
Keywords: palliative care; pediatrics; music therapy
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cognitively impaired children (Experimental): This is a single-group study; all participants will be offered the songwriting intervention.
  Interventions: Behavioral: Songwriting with licensed music therapist

INTERVENTIONS:
Behavioral: Songwriting with licensed music therapist — Song selected by parent-child dyad with recordings of physiologic components (i.e. heartbeat, breathing)

SUMMARY:
This study evaluates the feasibility and efficacy of a family-centered songwriting intervention for cognitively-impaired children referred to a palliative care service.

DETAILED DESCRIPTION:
Music-based interventions have previously been shown to reduce psychological distress in children with life-threatening conditions. However, children with cognitive impairment are frequently excluded from these studies. Our study will evaluate the efficacy a family-centered songwriting intervention for the following outcomes: child psychological and physical symptoms, parent psychological distress, and family environment.

Following recruitment, parent-child dyads will undergo 4 sessions with a licensed music therapist (anticipated to last 1 hour each). During these sessions, families and their children will select a song and engage in a songwriting process which includes various physiologic sounds from the child (i.e. heart rate, breathing). At the conclusion of these four sessions, a music DVD will be produced and delivered to the family.

ELIGIBILITY:
Inclusion Criteria:

* children ages 7-17 years
* cognitive impairment (T-score of 40 or below on the PROMIS Parent-Proxy Cognitive Function)
* receiving palliative/complex care
* progressively declining disease
* ability to hear.
* parents 18 years of age and older
* parent without cognitive impairment
* parent able to speak/understand English

Exclusion Criteria:

- None

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Intervention feasibility and recruitment log | throughout study completion, an average of 1 year
  Number of enrolled participants who complete all phases of study

SECONDARY OUTCOMES:
Parent Proxy Sleep Disturbance Short Form | Will be obtained at Time 1 (baseline, at recruitment) and at Time 2 (at completion of intervention, estimated at 3-4weeks following baseline)
  Parent-proxy measures of pediatric sleep disturbance. Scores range from 1 to 5; high scores indicate presence of disordered sleep symptoms, while low scores indicate absence of disordered sleep symptoms.
Parent Proxy Physical Stress Experiences | Will be obtained at Time 1 (baseline, at recruitment) and at Time 2 (at completion of intervention, estimated at 3-4weeks following baseline)
  Parent-proxy measures of pediatric physical stress. Includes eight Likert-scale questions. Scores range from 1 to 5; high scores indicate greater burden of physical stress experiences while low scores indicate lower likelihood of physical stress experiences.
Parent Proxy Psychological Stress Experiences | Will be obtained at Time 1 (baseline, at recruitment) and at Time 2 (at completion of intervention, estimated at 3-4weeks following baseline)
  Parent-proxy measures of pediatric psychological stress. Includes eight questions; scores range from 1 to five; high scores indicate higher level of psychological stress while low scores indicate lower levels of psychological stress.
Parent Proxy Anxiety | Will be obtained at Time 1 (baseline, at recruitment) and at Time 2 (at completion of intervention, estimated at 3-4weeks following baseline)
  Parent-proxy measures of pediatric anxiety. Includes eight Likert-scale questions with scores ranging from 1 to 5. High scores indicate more frequent child anxiety symptoms while low scores indicate less frequent child anxiety symptoms.
Parent Proxy Depressive Symptoms | Will be obtained at Time 1 (baseline, at recruitment) and at Time 2 (at completion of intervention, estimated at 3-4weeks following baseline)
  Parent-proxy measures of pediatric depressive symptoms. Includes six Likert-scale questions with scores ranging from 1-5. High scores indicate more frequent symptoms of pediatric depression, low scores indicate less frequent pediatric depressive symptoms.
Family Relationships | Will be obtained at Time 1 (baseline, at recruitment) and at Time 2 (at completion of intervention, estimated at 3-4weeks following baseline)
  Parent-proxy measures of family relationships symptoms. Includes eight Likert-scale questions which ranges from 1 to 5. High scores indicate higher family functioning and bonding while low scores indicate lower levels of family functioning and bonding.
Parent Anxiety | Will be obtained at Time 1 (baseline, at recruitment), at Time 2 (at completion of intervention, estimated at 3-4weeks following baseline), and at Time 3 (one month following death of child, if death of child occurs during study period.)
  Measure of parental anxiety symptoms. Includes eight Likert-scale questions with scores ranging from 1 to 5. Higher scores indicate elevation in parental anxiety while lower scores indicate lower levels of parental anxiety.
Parent Sleep Disturbance | Will be obtained at Time 1 (baseline, at recruitment), at Time 2 (at completion of intervention, estimated at 3-4weeks following baseline), and at Time 3 (one month following death of child, if death of child occurs during study period.)
  Measure of parental sleep disturbance. Includes four Likert-scale questions which range from 1 to 5. High scores indicate higher levels of disordered sleep while low scores indicate lower levels of disordered sleep.
Parental Perceived Stress (NIH Toolbox) | Will be obtained at Time 1 (baseline, at recruitment), at Time 2 (at completion of intervention, estimated at 3-4weeks following baseline), and at Time 3 (one month following death of child, if death of child occurs during study period.)
  Measure of parental perception of stress. Includes ten Likert-scale questions with scores ranging from 1 to 5. Higher scores indicate greater levels of parental perceived stress, while lower scores indicate lower levels of parental perceived stress.
Parent Satisfaction | Will be obtained at Time 2 (at completion of intervention, estimated at 3-4weeks following baseline), and at Time 3 (one month following death of child, if death of child occurs during study period.)
  Parents report satisfaction with songwriting intervention with qualitative responses.
Change in cortisol levels | Before and after each songwriting intervention session throughout study completion, an average of 1 year
  Salivary cortisol obtained from parent and child buccal swabs.

CONTACTS AND LOCATIONS:
Overall Officials: Terrah Akard, PhD, RN, Principal Investigator — Vanderbilt University
Locations (1):
- Monroe Carell, Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No